CLINICAL TRIAL: NCT07054567
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of BL-B01D1 + Pembrolizumab Dual Therapy With or Without Bevacizumab (BL-B01D1 + Pembrolizumab ± Bevacizumab) in Patients With Recurrent or Metastatic Cervical Cancer and Endometrial Cancer
Brief Title: A Study of BL-B01D1 + Pembrolizumab ± Bevacizumab in Patients With Recurrent or Metastatic Cervical Cancer and Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-204-11
Record Dates: First submitted 2025-06-20; First posted 2025-07-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — pembrolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 + pembrolizumab ± bevacizumab (Experimental): Participants receive BL-B01D1 + pembrolizumab ± bevacizumab in the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-B01D1; Drug: Pembrolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: Pembrolizumab — Administration by intravenous infusion for a cycle of 3 weeks.
Drug: Bevacizumab — Administration for a cycle of 3 weeks.

SUMMARY:
This Phase II study is a clinical trial to evaluate the efficacy and safety of BL-B01D1 + pembrolizumab dual therapy with or without bevacizumab (BL-B01D1 + pembrolizumab ± bevacizumab) in patients with recurrent or metastatic cervical cancer and endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily participates in this study and signs the informed consent form;
2. Age ≥18 years and ≤75 years;
3. Expected survival time ≥3 months;
4. ECOG performance status score of 0-1;
5. Patients with recurrent or metastatic cervical cancer or endometrial cancer confirmed by histopathology and/or cytology;
6. Archived tumor tissue samples from the primary or metastatic lesions within the past 3 years must be provided for PD-L1 and other testing;
7. Must have at least one measurable lesion as defined by RECIST v1.1;
8. Organ function levels must meet the requirements;
9. Toxicities from prior anti-tumor therapy must have recovered to ≤ Grade 1 as defined by NCI-CTCAE v5.0;
10. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, and the serum or urine pregnancy test must be negative. Patients must not be lactating. All enrolled patients must use adequate barrier contraception throughout the treatment period and for 6 months after treatment ends.

Exclusion Criteria:

1. Previously received ADC drugs with topoisomerase I inhibitors as the toxin or targeting EGFR and/or HER3;
2. Received chemotherapy, biological therapy, or immunotherapy within 4 weeks or 5 half-lives (whichever is shorter) before the first dose;
3. For Stage II (excluding Cohort 1), subjects who have previously received systemic anti-tumor therapy;
4. Prior immunotherapy resulting in ≥ Grade 3 irAE or ≥ Grade 2 immune-related myocarditis;
5. Used immunomodulatory drugs within 14 days before the first dose of the study drug;
6. Required systemic corticosteroid therapy within 2 weeks before the first dose of the study drug;
7. History of severe cardiovascular or cerebrovascular diseases;
8. Active autoimmune or inflammatory diseases;
9. Other malignancies that progressed or required treatment within 3 years before the first dose;
10. History of ILD/pneumonitis requiring steroid treatment, or current ILD/active pneumonitis;
11. Poorly controlled hypertension (requiring ≥ 2 antihypertensive medications);
12. Poorly controlled diabetes;
13. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
14. Active central nervous system metastases;
15. Patients with significant serous cavity effusion, symptomatic effusion, or poorly controlled effusion;
16. History of allergy to recombinant humanized antibodies or any excipients of the investigational drug;
17. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
18. Positive for HIV antibody, active tuberculosis, active hepatitis B virus (HBV) infection, or active hepatitis C virus (HCV) infection;
19. Active infection requiring systemic treatment;
20. Participation in another clinical trial within 4 weeks before the first dose;
21. Imaging shows tumor invasion or encasement of major abdominal, thoracic, cervical, or pharyngeal blood vessels;
22. Presence of severe unhealed wounds, ulcers, or fractures within 4 weeks before signing informed consent;
23. Clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing informed consent;
24. Planned or received live vaccines within 28 days before randomization;
25. History of severe neurological or psychiatric disorders;
26. Other conditions deemed by the investigator as unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 24 months
  Objective response rate (ORR) is defined as the number of CR and PR in the treatment and control groups divided by the number of that group in the full analysis set (FAS).
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of BL-B01D1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  Progression-free survival (PFS) as assessed by BICR is defined as the time between the date subjects are randomized and the first observation of disease progression (based on BICR's image-based assessment) or death.
Disease Control Rate (DCR) | Up to approximately 24 months
  Disease Control Rate (DCR) : Percentage of all randomized subjects who rated the best overall response (BOR) as complete response (CR), partial response (PR), and disease stabilization (SD) according to RECIST 1.1 criteria.
Duration of Response (DOR) | Up to approximately 24 months
  Duration of Response (DOR) : defined as the period from the date when tumor response is first recorded to the date when objective tumor progression is first recorded or the date of death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-B01D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-B01D1.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China